CLINICAL TRIAL: NCT05785026
Title: Effectiveness and Mechanisms of Menthol Inhalation for the Relief of Dyspnea in Health and COPD
Brief Title: Menthol for Dyspnea Relief in Health and COPD
Acronym: MENTHODYSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Daniel Langer, Assistant Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: S66762
Record Dates: First submitted 2023-02-07; First posted 2023-03-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Dyspnea; Chronic Obstructive Pulmonary Disease
Keywords: Menthol
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- WP 1a (Experimental): Menthol inhalation during resistive loaded breathing trials in healthy participants.
  Interventions: Other: Menthol inhalation
- WP 1b (Placebo Comparator): Strawberry scent during resistive loaded breathing trials in healthy participants.
  Interventions: Other: Strawberry scent
- WP 2a (Experimental): Menthol inhalation during cycle exercise in healthy participants.
  Interventions: Other: Menthol inhalation
- WP 2b (Placebo Comparator): Strawberry scent during cycle exercise in healthy participants.
  Interventions: Other: Strawberry scent
- WP 3a (Experimental): Menthol inhalation during resting breathing in dyspneic COPD participants.
  Interventions: Other: Menthol inhalation
- WP 3b (Placebo Comparator): Strawberry scent during resting breathing in dyspneic COPD participants.
  Interventions: Other: Strawberry scent
- WP 3c (No Intervention): Resting breathing in dyspneic COPD participants.
- WP 4a (Experimental): Menthol inhalation during cycle exercise in COPD participants.
  Interventions: Other: Menthol inhalation
- WP 4b (Placebo Comparator): Strawberry scent during cycle exercise in COPD participants.
  Interventions: Other: Strawberry scent
- WP 5a (Experimental): Menthol inhalation and facial airflow during cycle exercise in COPD participants
  Interventions: Other: Menthol inhalation and facial airflow
- WP 5b (Placebo Comparator): Strawberry inhalation and airflow to leg during cycle exercise in COPD participants
  Interventions: Other: Strawberry scent and airflow to leg
- WP 5c (Placebo Comparator): Menthol inhalation and airflow to leg during cycle exercise in COPD patients
  Interventions: Other: Menthol inhalation and airflow to leg
- WP 5d (Placebo Comparator): Strawberry inhalation and facial airflow during cycle exercise in COPD patients
  Interventions: Other: Strawberry inhalation and facial airflow

INTERVENTIONS:
Other: Menthol inhalation — 300 milligrams of L-menthol will be deposited on to a cellulose swab and secured inside the lower portion of a sealed facemask.
  Arms: WP 1a; WP 2a; WP 3a; WP 4a
Other: Strawberry scent — 600 microliters of 100% natural strawberry flavoring will be deposited onto on to a cellulose swab and secured inside the lower portion of a sealed facemask.
  Arms: WP 1b; WP 2b; WP 3b; WP 4b
Other: Menthol inhalation and facial airflow — Menthol will be administered using a noseplug and facial airflow will be applied with a tabletop fan.
  Arms: WP 5a
Other: Strawberry scent and airflow to leg — Strawberry will be administered using a noseplug and airflow to the leg will be applied with a tabletop fan.
  Arms: WP 5b
Other: Menthol inhalation and airflow to leg — Menthol will be administered using a noseplug and airflow to the leg will be applied with a tabletop fan.
  Arms: WP 5c
Other: Strawberry inhalation and facial airflow — Strawberry will be administered using a noseplug and facial airflow will be applied with a tabletop fan.
  Arms: WP 5d

SUMMARY:
Menthol inhalation (MI) is a novel and promising treatment option for acute relief of dyspnea, however, the underlying ventilatory and/or neural related mechanisms for this relief in symptoms remain unknown. The overall aim of this research project is to systematically examine the mechanisms of dyspnea relief from MI in healthy individuals and those with COPD.

DETAILED DESCRIPTION:
The project is structured in 5 work packages (WP), each including a different sample of healthy volunteers (WP1, 2) or patients with COPD (WP3, 4, 5), respectively with a 1:1 female/male ratio in each WP. Each WP will be single-blind, placebo-controlled cross-over trial to investigate the effects of MI compared to placebo in healthy volunteers during resistive loaded breathing (WP1), in healthy volunteers during cycling exercise (WP2), in people with COPD who have dyspnea at rest (WP3), and in people with COPD during cycling exercise (WP4, 5).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years of age or older
* Able to speak, read, and write Dutch or English
* Normal pulmonary function: forced expiratory volume in 1 second (FEV1) to forced vital capacity ratio>0.70; FEV1≥80%predicted (WP1 and 2 only)
* Non-smoker or former smokers (smoke-free ≥12 months prior to enrolment) (WP1 and 2 only)
* Clinically stable COPD (based on clinical judgment of the study physician that have not had exacerbations requiring escalation of medical therapy (i.e., short course of oral corticosteroids or antibiotics) within the preceding 14 days (WP3 and 4 only)

Exclusion Criteria:

* Contraindication to exercise testing (e.g., significant cardiovascular, musculoskeletal, neurological disease; see Table 4 from ERS/ATS consensus statement)
* Significant pulmonary or extra-pulmonary disease that, based on clinical assessment, could influence dyspnea and/or impair exercise capacity (with the exception of COPD in WP3 and 4)
* Body mass index <18.5 or >35 kg/m2
* An ulcer or tumor in the esophagus, a nasal septum deviation, or recent nasopharyngeal surgery
* Severe facial trauma including cribriform plate disruption (bone separating brain from nasal cavity)
* Allergies to latex and sensitivities to local anesthetics
* Inability to give informed consent, including those with significant cognitive impairment
* Alcohol consumption within 12 hours of study visit
* Current smoker*
* History of early menopause (age <45 years)
* Pregnancy or desire to become pregnant while in trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Difference in respiratory-related evoked potentials (RREP) with menthol vs. strawberry. | 1 week
  RREPs will be measured using an electroencephalogram (EEG) sensor cap connected to a high-density 129 channel EEG system during breathing trials and exercise tests. Inspiration will briefly be interrupted for 150 milliseconds every two to six breaths by activation of the occluder, which induces the RREP in the EEG signal.

OTHER OUTCOMES:
Difference in diaphragmatic electromyography with menthol vs. strawberry. | 1 week
  Diaphragmatic electromyography will be measured using a multi-pair electrode catheter during breathing trials and exercise tests. and used as an index of neural respiratory drive.
Difference in dyspnea with menthol vs. strawberry (+ facial airflow or airflow to leg in WP5). | 1 week
  Dyspnea ratings will be measured using the Borg 0-10 category ratio scale and will be assessed at the end of each 5-minute breathing trial (WP1 and 3), and at baseline, every minute during (WP4,5) or halfway through the test (WP2), and at peak of each cycle exercise test. 0 represents no dyspnea at all and then 10 the most maximal dyspnea ever experienced or could be imagined experiencing.
Difference in the rate of perceived inspiratory airflow. | 1 week
  Participants will be asked: "In which of the four conditions did your airflow feel easier when breathing in?" at the end of each study visit.
Perception of a cooling sensation. | 1 week
  Participants will be asked: "In which of the four conditions did you feel a fresh or cooling sensation when breathing in?" at the end of each study visit.
Difference in activation of extra-diaphragmatic inspiratory muscles with menthol vs. strawberry. | 1 week
  Activation of extra-diaphragmatic inspiratory muscles will be measured using bipolar surface electrodes during breathing trials (WP3) and exercise testing (WP4).
Difference in the cardiorespiratory responses to exercise with menthol vs. strawberry. | 1 week
  Cardiorespiratory responses to exercise will be measured on a breath-by-breath basis using a commercially available cardiopulmonary testing system during exercise testing.
Difference in respiratory pressures with menthol vs. strawberry. | 1 week
  Respiratory pressures will be measured using esophageal and gastric balloons during breathing trials and exercise testing.
Difference in leg discomfort ratings with menthol vs. strawberry (+facial airflow or airflow to leg in WP5). | 1 week
  Leg discomfort will be measured using the Borg 0-10 category ratio scale at baseline, every minute during (WP4, 5) or halfway through the test (WP2), and at peak of each cycle exercise test. 0 represents no leg discomfort at all and then 10 the most maximal leg discomfort ever experienced or could be imagined experiencing.
Difference in exercise endurance time with menthol vs. strawberry (+ facial airflow or airflow to leg in WP5). | 1 week
  Exercise endurance time will be measured during submaximal constant load cycle exercise testing (WP4, 5).
Difference in the reasons for stopping exercise with menthol vs. strawberry (+facial airflow or airflow to leg in WP5). | 1 week
  Participants will be asked to give their reasons for stopping (e.g., "breathing discomfort," "leg discomfort," "a combination of breathing and leg discomfort," or "other") and attributing a percentage to each of breathing discomfort and leg discomfort to total 100 (WP 2, 4 and 5).
Difference in ratings of affective state on the dimensions of valence and arousal with menthol vs. strawberry (+ facial airflow or airflow to leg in WP5). | 1 week
  Dimensions of valence and arousal will be measured using the 9-point Self-Assessment Manikin scale for valence (1 -"unpleasant" to 9 -"pleasant") and arousal (1-"calm" to 9-"aroused") at the end of each breathing trial (WP 1 and 3) and at peak exercise (WP 2, 4 and 5).
Difference in the Neural Drive to Breathe (P0.1) | 1 week
  The neural drive to breathe will be measured using airway occlusion pressure (P0.1), evoked by inspiratory occlusions delivered during the test (WP1 and 2).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langer, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schaeffer MR, Vanden Bossche L, Beckers K, Verbeke K, Janssens W, Jensen D, Arnold JI, von Leupoldt A, Langer D. Inhaled Menthol for Dyspnea Relief During Cycle Exercise in COPD: A Randomized Trial. Chest. 2025 Aug;168(2):390-401. doi: 10.1016/j.chest.2025.03.002. Epub 2025 Mar 13. PMID 40088943